CLINICAL TRIAL: NCT00530764
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Dose-range Exploration Study of Sativex® in Relieving Pain in Patients With Advanced Cancer, Who Experience Inadequate Analgesia During Optimized Chronic Opioid Therapy.
Brief Title: A Study of Sativex® for Pain Relief in Patients With Advanced Malignancy.
Acronym: SPRAY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWCA0701
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Palliative Care; Pain; Cancer
Keywords: Pain; Cancer; Palliative
MeSH Terms: conditions — Pain; Neoplasms | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sativex Low Dose (Experimental): Range of 1 to 4 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 10.8mg THC and 10mg CBD.
  Interventions: Drug: Sativex Low Dose
- Sativex Medium Dose (Experimental): Range of 6 to 10 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 27mg THC and 25mg CBD.
  Interventions: Drug: Sativex Medium Dose
- Sativex High Dose (Experimental): Range of 11 to 16 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 43.2mg THC and 40mg CBD.
  Interventions: Drug: Sativex High Dose
- Placebo (No Intervention): Range of 1-16 sprays per day of placebo spray.

INTERVENTIONS:
Drug: Sativex Low Dose — Range of 1 to 4 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 10.8mg THC and 10mg CBD.
  Other Names: GW-1000-02
  Arms: Sativex Low Dose
Drug: Sativex Medium Dose — Range of 6 to 10 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 27mg THC and 25mg CBD.
  Other Names: GW-1000-02
  Arms: Sativex Medium Dose
Drug: Sativex High Dose — Range of 11 to 16 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 43.2mg THC and 40mg CBD.
  Other Names: GW-1000-02
  Arms: Sativex High Dose

SUMMARY:
The purpose of this study is to determine the effective dose range and to demonstrate a non-effective dose range of Sativex in patients with advanced cancer, who experience inadequate pain relief even though they are on optimized chronic opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient has advanced active cancer for which there is no known curative therapy.
* The patient is able (in the investigators opinion) and willing to comply with all study requirements.
* The patient has a clinical diagnosis of cancer related pain, which is not wholly alleviated with their current opioid treatment.
* The patient is receiving a sustained release (SR) fixed dose of opioid therapy (excluding Methadone). N.B. The opiate therapy must be Step III according to the World Health Organization (WHO) analgesic ladder.
* The patient is willing to continue to take their regular daily baseline opioid regimen (SR) at the same dose, throughout the duration of study.

Exclusion Criteria:

* The patient should be excluded from entering study if they have received or are due to receive during the study period; chemotherapy, hormone therapy or radiotherapy, which, in the opinion of the investigator will affect their pain.
* Any history or immediate family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Any known or suspected history of a diagnosed dependence disorder, current heavy alcohol consumption, current use of an illicit drug or current non prescribed use of any prescription drug.
* The patient has poorly controlled epilepsy or recurrent seizures (i.e. at least one year since last seizure).
* The patient has experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or has a cardiac disorder that, in the opinion of the investigator would put the patient at risk of a clinically relevant arrhythmia or myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (23):
  - Cancer Care Center of Tuscaloosa, Tuscaloosa, Alabama
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - Office of Dr. Ronald Yanagihara, Gilroy, California
  - University of California San Diego, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Center of Hope for Cancer and Blood Disorders, Riverdale, Georgia
  - Louisiana Research Associates, New Orleans, Louisiana
  - The Center for Clinical Research - Washington County Hospital, Hagerstown, Maryland
  - Capital Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - A & A Pain Institute of St. Louis, St Louis, Missouri
  - Office of Donald H. Berdeaux MD, Great Falls, Montana
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Metropolitan Hospital Center, New York, New York
  - Four Seasons Hospice & Pallative Care, Flat Rock, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Lone Star Oncology, Austin, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Belgium (3):
  - Jules Bordet Institute, Brussels
  - CHU Charleroi (Hôpital civil de Charleroi), Charleroi
  - UZ Leuven - Algologisch Centrum Anesthesiologie, Pellenberg
- Canada (2):
  - Vancouver Health Research Center, Victoria, British Columbia
  - Jewish General Hospital, Montreal, Quebec
- Chile (2):
  - Instituto Radio-oncológico Santiago (INRAD), Santiago
  - Clínica Ciudad del Mar, Viña del Mar
- Czechia (9):
  - Ambulance pro lécbu bolesti, ARO, Benešov
  - Ambulance pro lécbu bolesti, České Budějovice
  - Nemocnice Ceské Budejovice, České Budějovice
  - FN Hradec Králové - Klinika onkologie a radioterapie, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - FN a LF UP Olomouc - Ambulance pro lécbu bolesti, Olomouc
  - AR klinika FN Plzen -Ambulance pro lécbu bolesti, Pilsen
  - Fakultní nemocnice Na Bulovce, Praha 8 - Liben
  - ARO, Krajská zdravotni, K.Z. a.s, Nemocnice, Teplice
- Docrates Clinic, Helsinki, Finland
- France (2):
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Praticien hospitalier, Tarbes
- Germany (4):
  - RWTH Aachen Universität, Aachen
  - Schmerz- und Palliativzentrum Göppingen, Göppingen
  - St.-Marien-Hospital Lunen, Lünen
  - Schmeiz - u Pallielivzendium Wiesbaden, Wiesbaden
- India (13):
  - Yashoda Hospital, Andhra Pradesh
  - Bangalore Institute of Oncology, Bangalore
  - CBCC- Apollo Hospital, Gandhinagar
  - Apollo Hospital, Hyderabaad
  - Indo-American Cancer Institute and Research Center, Hyderabaad
  - Bhagwaan Mahaveer Cancer Hospital and Research Centre, Jaipur
  - CHL - Apollo Hospitals, Madhya Pradesh
  - Jawaharlal Nehru Cancer Hospital, Madhya Pradesh
  - Meenakshi Mission Hospital & Research Centre, Madurai
  - All India Institute of Medical Sciences, New Delhi
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
  - Deenanath Mangeshkar Hospital and Research Center, Pune
  - Seroc Cancer Center, Rajasthan
- Italy (2):
  - Regina Elana Cancer Institute, Rome
  - Dir. S.C.D.U. Psicologia Clinica ed Oncologica, Turin
- Mexico (2):
  - Hospital Aranda de la Parra, León
  - Htal Ángeles de Pedregal, Mexico City
- Poland (8):
  - Beskidzkie Centrum Onkologii im. Jana Pawla, Bielsko-Biala
  - Poradnia Leczenia Bolu, Edyty Jakubow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Gdansk
  - NZOZ Hospicjum Milosierdzia Bozego, Gliwice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wielkopolskie Centrum Onkologii, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej, Tychy
  - Centrum Onkologii - Instytut im. M. Sklodowskiej - Curie, Warsaw
- Romania (12):
  - Spitalul Judetean de Urgenta "Constantin Opris", Baia Mare, Maramures
  - Spitalul Judetean de Urgenta Braila, Braila, Jud. Braila
  - Hospice "Casa Sperantei", Brasov
  - Spitalul Universitar de Urgenta Elias, Bucharest
  - S.C. IanuliMed S.R.L. Oncologie Medicala, Bucharest
  - Policnica Orizont-Oncologie Medicala, Craiova
  - District Hospital Dr. Alexandru Simionescu, Hunedoara
  - Centrul de Oncologie Medicala, Iași
  - Spitalul Municipal Onesti, Onesti, Jud. Bacau
  - Spitalul Municipal Ploiesti, Ploieşti
  - Spitalul Clinic Judetean Sibiu Oncologie, Sibiu
  - Spitalul Judetean de Urgenta "Sf. Ioan cel Nou", Suceava
- South Africa (7):
  - Medi Clinic, Bloemfontein
  - Pain Clinic, Cape Town
  - Dr. Pirjol & Szpak Inc., eManzimtoti
  - Pretoria Urology Research Unit, Hatfield, Pretoria
  - Trialtech Research - Embassy Drive Medical Centre, Hatfield, Pretoria
  - Oncology/Haematology Dept Research Unit, Kimberley
  - Eastleigh Breast Cancer Center, Lynnwood
- Spain (8):
  - Hospital Virgen del Mar, Almería
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - HU Puerta del Mar, Oncologia, Cadiz
  - Hospital Universitario de Bellvitge, Feixa, Llarga, Sn
  - Hospital Univ. Virgen de las Nieves, Granada
  - Hospital de la Rioja, Logroño
  - Hospital Los Montalvos, Salamanca
- United Kingdom (12):
  - Basingstoke & North Hampshire NHS Foundation Trust, Basingstoke
  - West Suffolk Hospital, Bury St Edmunds
  - Fairfield General Hospital, Bury, Lancashire
  - Edinburgh Cancer Research Centre (CRUK), Edinburgh
  - James Paget Hospital, Gorleston on Sea, Norfolk
  - International Observatory on End of Life Care, Lancaster
  - St Bartholomew's Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Marie Curie Hospice Holme Tower, Penarth
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Weston Area Health Trust, Weston-super-Mare
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Result] Portenoy RK, Ganae-Motan ED, Allende S, Yanagihara R, Shaiova L, Weinstein S, McQuade R, Wright S, Fallon MT. Nabiximols for opioid-treated cancer patients with poorly-controlled chronic pain: a randomized, placebo-controlled, graded-dose trial. J Pain. 2012 May;13(5):438-49. doi: 10.1016/j.jpain.2012.01.003. Epub 2012 Apr 5. PMID 22483680

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex High Dose Group: Range of 11 to 16 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 43.2mg THC and 40mg CBD.
- Sativex Medium Dose Group: Range of 6 to 10 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 27mg THC and 25mg CBD.
- Sativex Low Dose Group: Range of 1 to 4 sprays per day. Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). Thus maximum daily dose is 10.8mg THC and 10mg CBD.
Period: Overall Study
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Started | 90 | 88 | 91 | 91
Completed | 59 | 67 | 71 | 66
Not Completed | 31 | 21 | 20 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo | Total
Number analyzed (Participants) | 90 | 88 | 91 | 91 | 360
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (11.2) | 59 (31.1) | 59 (12.3) | 56 (12.2) | 58 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 46 | 47 | 174
  Male | 48 | 49 | 45 | 44 | 186

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least 30% Improvement in Numerical Rating Scale (NRS) Average Pain Score From Baseline
Description: A positive 30% pain response is defined as a reduction of at least 30% in the mean NRS average pain score from baseline to week 5 (last 3 days). The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to cancer. The average pain NRS was completed at the same time each day, i.e. bedtime in the evening.
Time Frame: 5 Weeks: Baseline (first 3 days) - Week 5 (last 3 days)
Measure: Number; unit: Participants
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 90 | 87 | 91 | 91
Participants | 22 [0.46 to 1.76] | 26 [0.62 to 2.28] | 30 [0.72 to 2.60] | 24
Statistical Analysis 1: Comparison: Sativex Low Dose Group vs Placebo; The proportions of responders were compared between the treatment groups using logistic regression with region and treatment groups as factors. The null hypothesis was that there was no difference between each of the Sativex treatment groups and placebo. The estimated response rates, odds ratios, 95% CIs for the odds ratios and p-values were presented; Test type: Superiority or Other; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.72 to 2.60]
Statistical Analysis 2: Comparison: Sativex High Dose Group vs Placebo; As for Sativex Low dose versus placebo; Test type: Superiority or Other; p = 0.62, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.46 to 1.76]
Statistical Analysis 3: Comparison: Sativex Medium Dose Group vs Placebo; As for Sativex Low dose versus placebo; Test type: Superiority or Other; p = 0.61, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.62 to 2.28]

2. Secondary Outcome: Change in Cumulative Average Pain Response Curves
Description: The cumulative response to treatment is the percentage changes from baseline in the mean NRS pain score as defined as the 30% response.
  The pain NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to cancer.
Time Frame: Baseline to end of treatment (Week 5)
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 89 | 87 | 89 | 91
Percent Change | -13 [-30 to 6] | -20 [-40 to -6] | -20 [-48 to -8] | -10 [-33 to 5]
Statistical Analysis 1: Comparison: Sativex Low Dose Group vs Placebo; Each of the active treatment groups were compared with placebo using pairwise Wilcoxon rank-sum tests. The Hodges-Lehmann estimates and 95% CI for the median differences were also presented; Test type: Superiority or Other; p = 0.0077, Wilcoxon rank sum tests; Median Difference (Final Values) = -12.5, 95% CI 2-sided [-21.35 to -3.33]
Statistical Analysis 2: Comparison: Sativex High Dose Group vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.67, Wilcoxin rank sum test; Median Difference (Final Values) = -1.97, 95% CI 2-sided [-11.04 to 7.14]
Statistical Analysis 3: Comparison: Sativex Medium Dose Group vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.039, Wilcoxin rank sum test; Median Difference (Final Values) = -8.75, 95% CI 2-sided [-17.14 to 0.00]

3. Secondary Outcome: Change in Mean Daily NRS Pain Score (Average Pain).
Description: The average pain NRS was complete at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to cancer. A negative value indicates an improvement in pain score from baseline.
Time Frame: 5 Weeks: Baseline (first 3 days) - End of Treatment (last 3 days of week 5)
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Sativex High Dose | Sativex Medium Dose | Sativex Low Dose | Placebo
Number analyzed (Participants) | 89 | 87 | 89 | 91
Points on scale | -0.9 (1.9) [-6.3 to 2.3] | -1.2 (1.7) [-7.3 to 5.7] | -1.6 (2.1) [-8.0 to 3.3] | -0.8 (1.8) [-6.0 to 3.7]
Statistical Analysis 1: Comparison: Sativex Low Dose vs Placebo; The change in mean pain NRS score (average pain) was analyzed using analysis of covariance (ANCOVA) with the baseline value as a covariate and region and treatment group as factors; Test type: Superiority or Other; p = 0.006, ANCOVA; Estimated treatment effect = -0.75, 95% CI 2-sided [-1.28 to -0.22]
Statistical Analysis 2: Comparison: Sativex High Dose vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.75, ANCOVA; Estimated treatment effect = -0.09, 95% CI 2-sided [-0.62 to 0.44]
Statistical Analysis 3: Comparison: Sativex Medium Dose vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.19, ANCOVA; Estimated treatment effect = -0.36, 95% CI 2-sided [-0.89 to 0.18]

4. Secondary Outcome: Change in Mean Daily NRS Pain Score (Worst Pain).
Description: The worst pain NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your worst pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to cancer. A negative value indicates an improvement in worst pain score from baseline.
Time Frame: 5 Weeks: Baseline (first 3 days) - End of Treatment (last 3 days of week 5)
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Sativex High Dose | Sativex Medium Dose | Sativex Low Dose | Placebo
Number analyzed (Participants) | 89 | 87 | 89 | 91
Points on scale | -1.0 (1.9) | -1.2 (1.8) | -1.6 (2.2) | -0.9 (2.0)
Statistical Analysis 1: Comparison: Sativex Low Dose vs Placebo; The change in mean pain NRS score (worst pain) was analyzed using ANCOVA with the baseline value as a covariate and region and treatment group as factors; Test type: Superiority or Other; p = 0.011, ANCOVA; Estimated treatment effect = -0.73, 95% CI 2-sided [-1.30 to -0.17]
Statistical Analysis 2: Comparison: Sativex High Dose vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.14, ANCOVA; Estimated treatment effect = -0.35, 95% CI 2-sided [-0.81 to 0.11]
Statistical Analysis 3: Comparison: Sativex Medium Dose vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.40, ANCOVA; Estimated Treatment Effect = -0.24, 95% CI 2-sided [-0.81 to 0.32]

5. Secondary Outcome: Change in Sleep Disruption NRS
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: 5 Weeks: Baseline - End of Treatment (Last 3 days of Week 5)
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 89 | 87 | 89 | 91
Points on scale | -0.7 (2.1) [-1.45 to -0.31] | -0.9 (2.1) [-1.45 to -0.31] | -1.5 (2.1) [-1.45 to -0.31] | -0.8 (2.2)
Statistical Analysis 1: Comparison: Sativex Low Dose Group vs Placebo; The change in mean sleep disturbance NRS score was analyzed using ANCOVA with the baseline value as a covariate and region and treatment group as factors; Test type: Superiority or Other; p = 0.003, ANCOVA; Estimated Treatment Effect = -0.88, 95% CI 2-sided [-1.45 to -0.31]
Statistical Analysis 2: Comparison: Sativex High Dose Group vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.78, ANCOVA; Estimated Treatment Effect = -0.08, 95% CI 2-sided [-0.65 to 0.49]
Statistical Analysis 3: Comparison: Sativex Medium Dose Group vs Placebo; As for Sativex low dose versus placebo; Test type: Superiority or Other; p = 0.26, ANCOVA; Estimated Treatment Effect = -0.33, 95% CI 2-sided [-0.90 to 0.24]

6. Secondary Outcome: Change in Brief Pain Inventory - Short Form (BPI-SF)
Description: The BPI-SF is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items(range 0-10). the minimum value is zero and maximum is 10. A higher score represents a poor outcome.
Time Frame: Baseline (Visit 2) and End of Treatment (End of Week 5 or premature termination)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 68 | 68 | 69 | 74
Score on scale | -1.0 (1.9) [.09 to .34] | -1.5 (1.6) [.09 to .34] | -1.3 (2.3) [.09 to .34] | -1.0 (1.9)

7. Secondary Outcome: Change in Patient Assessment of Constipation Quality of Life (PAC-QoL)
Description: The PAC-QoL questionnaire consists of 28 questions divided into the following areas: 4 questions on physical discomfort, 8 questions on psychosocial discomfort, 11 questions on worries/concerns and 5 questions on satisfaction. The PAC-QoL was completed at baseline and then at the end of treatment. An overall score (range 0-4) was calculated at each visit and the difference determined. A positive difference in score represents an improvement.
Time Frame: Baseline (Visit 2) and End of Treatment (Week 5 or premature termination)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 74
Score on scale | 0.0 (0.7) [-0.04 to 0.26] | -0.1 (0.5) [-0.04 to 0.26] | 0.0 (0.6) [-0.04 to 0.26] | -0.1 (0.6)

8. Secondary Outcome: Change in Patient Global Impression of Change - PGIC
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your pain due to cancer since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At Visit 2 (Baseline) patients wrote a brief description of their pain caused by cancer which was used at Week 5 to aid their memory regarding their symptoms at study start. For each of above markers the number of participants were reported.
Time Frame: End of Week 5
Measure: Number; unit: Participants
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 73 | 71 | 70 | 72
Participants
  Very much improved | 6 [0.46 to 1.49] | 6 [0.49 to 1.58] | 10 [0.77 to 2.53] | 9
  Much improved | 20 | 19 | 24 | 16
  Slightly improved | 25 | 26 | 19 | 28
  No change | 13 | 13 | 13 | 17
  Slightly worse | 6 | 5 | 3 | 1
  Much worse | 1 | 0 | 1 | 1
  Very much worse | 2 | 2 | 0 | 0

9. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS comprises of 10 questions that are completed by the patient to determine their depression level. The MADRS was completed at Visit 2 (Baseline) prior to receiving the study drug and at Visit 4 (Week 5 or premature termination). Each item is scored on a 0-6 scale , where 0=no sadness to 6=extreme and continuous gloom and despondency, and the MADRS score is the sum of the 10 item scores (range 0-60). The higher the score the more severe the depression.
Time Frame: Baseline and End of Treatment (Week 5 or premature termination)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Number analyzed (Participants) | 67 | 66 | 66 | 69
Score on scale | -0.4 (8.6) [0.38 to 3.74] | -1.0 (8.5) [0.38 to 3.74] | -1.1 (7.0) [0.38 to 3.74] | -2.9 (9.0)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring from the time of consent to post study follow up (Visit 5) i.e.9 weeks were collected. All deaths and serious adverse events (SAEs) occurring within 28 days of the final dose of study medication were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex High Dose Group | Sativex Medium Dose Group | Sativex Low Dose Group | Placebo
Serious Adverse Events (participants affected / at risk) | 28/90 | 18/87 | 35/91 | 23/91
Other Adverse Events (participants affected / at risk) | 82/90 | 73/87 | 68/91 | 69/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sativex High Dose Group (N=90) | Sativex Medium Dose Group (N=87) | Sativex Low Dose Group (N=91) | Placebo (N=91)
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2
Cardiac disorders (Cardiac disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 4 | 3 | 1 | 2
General Disorders (General disorders) | 4 | 1 | 4 | 2 — Any new unfavorable/unintended symptoms, worsening of condition that may/not be considered related to study medication.
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Infections and Infestations (Infections and infestations) | 2 | 5 | 4 | 2
Injury, Poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Investigations (Investigations) | 1 | 0 | 0 | 0
Metabolism and Nutrition disorders (Metabolism and nutrition disorders) | 3 | 1 | 1/87 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (Incl. Cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 12 | 26 | 15
Nervous system disorders (Nervous system disorders) | 3 | 1 | 1 | 0
Psychiatric disorders (Psychiatric disorders) | 2 | 1 | 1 | 0
Renal and urinary disorders (Renal and urinary disorders) | 4 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Vascular disorders (Vascular disorders) | 3 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sativex High Dose Group (N=90) | Sativex Medium Dose Group (N=87) | Sativex Low Dose Group (N=91) | Placebo (N=91)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 9 | 8 | 9 | 7
Cardiac disorders (Cardiac disorders) | 2 | 2 | 6 | 6
Ear and labyrinth disorders (Ear and labyrinth disorders) | 4 | 4 | 0 | 3
Eye disorders (Eye disorders) | 1 | 4 | 1 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 47 | 42 | 36 | 29
General Disorders (General disorders) | 24 | 18 | 18 | 20
Hepatobillary Disorders (Hepatobiliary disorders) | 2 | 1 | 0 | 0
Infections and Infestations (Infections and infestations) | 8 | 15 | 11/81 | 11
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 4
Investigations (Investigations) | 5 | 9 | 11 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 22 | 15 | 11 | 12
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 | 12 | 6 | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 12 | 26 | 14
Nervous system disorders (Nervous system disorders) | 44 | 39 | 26 | 20
Psychiatric disorders (Psychiatric disorders) | 23 | 14 | 13 | 13
Renal and urinary disorders (Renal and urinary disorders) | 8 | 4 | 4 | 6
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 11 | 6
Skin and subcuraneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 | 3 | 3 | 1
Surgical and medical procedures (Surgical and medical procedures) | 0 | 0 | 2 | 0
Vascular Disorders (Vascular disorders) | 4 | 3 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Policy:

GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications for example, manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.